CLINICAL TRIAL: NCT05122468
Title: The Use of a Connective Tissue Auto-graft in Combination With Either the Tunnel Technique or the Coronally Advanced Flap for the Treatment of Multiple Gingival Recession Defects. A Randomized Controlled Clinical Trial.
Brief Title: Tunnel vs. CAF for the Treatment of Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Jerian González-Febles, Principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.I. 16/504
Record Dates: First submitted 2021-05-03; First posted 2021-11-16 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The two intervention groups will be the CAF group (standard of care control) and Tunnel group (TUN, Test group). Two experienced clinicians (ML, or JG) will deliver treatment consisting of root coverage surgery using a coronally advanced flap in combination with a connective tissue graft (Control group), or a tunnel technique (Test group) in combination with a connective tissue graft.
  Follow-up of individual patients will be 6 months (to be extended to 3 years to observe differences in a long-term basis)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A connective tissue graft will be harvested from the palate as a free gingival graft, which will be de-epithelialized with a 15-c blade(Zucchelli et al. 2010) before opening of the opaque envelopes, which contains the allocation concealment. Afterwards, test or control procedure will be carried out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF group (Active Comparator): Coronally advanced flap in combination with a connective tissue graft.
  According to the technique(Zucchelli & De Sanctis 2000), this procedure consists of a rotated papilla, envelope flap. Intrasulcular incisions will be performed involving all the experimental units and at least one tooth mesial and distal to the experimental teeth. From the centre of rotation the incisions will be traced in a corono-apical direction toward the mesial and toward the distal extension of the flap.
  After the accurate initial incisions, the flap will be raised full thickness apical to the mucogingival junction (MGJ), exposing 1 to 2 mm of bone at the base of the recession/dehiscence defects.
  A linear mesio-distal incision will then be performed to cut the periosteum, releasing any muscular tension and allow a passive coronal positioning of the flap to cover the CEJ.
  Interventions: Procedure: Connective tissue Harvest and CAF
- Tunnel group (Experimental): Tunnel technique in combination with a connective tissue graft.
  When tunnelling procedures are applied, this technique consists of a supra-periosteal bed under a pedicle flap without any external incisions (Zabalegui et al. 1999). Afterwards, a connective tissue graft is placed and secured through the tunnel, covering the adjacent exposed roots.
  To create a tunnel at the buccal aspect of the gingiva, sulcular partial-thickness incisions are made by means of a micro-blade through each recession area, extending the split-thickness beyond the mucogingival junction (MGJ). The partial dissection plane is then extended laterally through the papillae between the treated teeth without separating them. This incision must also be extended 3 to 5 mm mesial and distal from the lateral teeth to allow space for the connective tissue graft.
  Interventions: Procedure: Connective tissue Harvest and Tunnel

INTERVENTIONS:
Procedure: Connective tissue Harvest and CAF — A connective tissue graft will be harvested from the palate as a free gingival graft, which will be de-epithelialized with a 15-c blade(Zucchelli et al. 2010) before opening of the opaque envelopes, which contains the allocation concealment. The dimensions of the graft achieve 3 to 5 mm mesial and distal from the lateral teeth with an ideal thickness about 1 to 1.5 mm. Donor tissue will be taken at premolar and molar level. In control sites, the graft will be adapted to cover each exposed root to the CEJ, and stabilized with either 6-0 resorbable sutures (with the knot placed under the papillary area) or a non-resorbable suture with the knot on the palatal side. For suturing of the graft, interrupted sutures or sling sutures (anchored to periosteum apical to the graft and hanging around the neck of the experimental teeth) may be used.
  Arms: CAF group
Procedure: Connective tissue Harvest and Tunnel — A connective tissue graft will be harvested from the palate as a free gingival graft, which will be de-epithelialized with a 15-c blade(Zucchelli et al. 2010) before opening of the opaque envelopes, which contains the allocation concealment. The dimensions of the graft achieve 3 to 5 mm mesial and distal from the lateral teeth with an ideal thickness about 1 to 1.5 mm. Donor tissue will be taken at premolar and molar level.
  In test sites, the graft should be slid through the tunnel. To accomplish the adequate position of the graft into the tunnel, 2 sutures are first placed, 1 at the most mesial and the other at the most distal aspect of the tunnel. The needles should pass underneath the tunnel and exit through the largest or most central gingival recession, the one through which the grafting tissue will be introduced. With these 2 sutures already inside the tunnel, the graft is bitten on both ends with vertical mattress sutures.
  Arms: Tunnel group

SUMMARY:
Many studies have compared the tunnel technique and coronally advanced flap in the treatment of single and multiple recessions. However, there is a lack of evidence that compared both techniques in combination with a connective tissue graft, for just multiple adjacent recessions. No technique is clearly superior to another in terms of complete root coverage (CRC), mean root coverage (MRC) and the gain of keratinized tissue height (KTH) when multiple recession coverage was evaluated. Moreover, as a connective tissue graft supposed to offer more stability in terms of complete root coverage in long-term basis, the main question should be aimed at the role of the sub-epithelial connective tissue graft, when it is used in combination with one technique or another. Hence, the hypothesis is focused on if the use of a connective tissue graft in combination with a tunnel technique would provide higher clinical outcomes and similar patient-based outcomes than its use in combination with the Coronally Advanced flap technique.

DETAILED DESCRIPTION:
Parallel group, clinical evaluator- and statistician-blinded, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

• Subjects with a minimum of two adjacent teeth and a maximum of four adjacent teeth with gingival recessions (at least one with a depth ≥ 3 mm) and requiring surgical intervention, without medical contraindications to elective surgery.

Exclusion Criteria:

* Presence of untreated periodontitis
* Persistence of uncorrected gingival trauma from tooth brushing
* Interdental attachment loss greater than 1 mm or furcation involvement in the teeth to be treated
* Presence of severe tooth malposition, rotation or clinically significant super-eruption
* Self-reported current smoking
* Presence of medical contraindications to elective surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Complete root coverage | 6 months
  The complete root coverage is defined as the percentage of cases that 100% of the recessions will be covered in their whole extension.

SECONDARY OUTCOMES:
Mean Root Coverage | 6 months
  The mean root coverage is the percentage of recession extension, which will be covered at 6 months after surgery.
Recession Reduction (RR) | 6 months
  It is described as the changes in recession measurements between baseline and 6 months post-operative. Recession is defined as position of the gingival margin. All included recessions will be measured with two methods:
  1. from the CEJ to the gingival margin
  2. from the incisal edge to the gingival margin All measures will be taken using as reference the most apical position of the gingival margin on the facial aspect of the tooth.
Probing pocket depth (PPD) | 6 months
  Depth of the gingival sulcus/pocket will be assessed on the mid-facial aspect of each tooth. The width of keratinized tissue will be assessed clinically, while attached gingival will be derived mathematically subtracting the width of keratinized gingiva and the depth of the sulcus/pocket.
Clinical attachment Gain | 6 months
  It is the change in clinical attachment levels between baseline and 6 Months post-opeartive. Clinical attachment level is defined as the sum of recession and probing pocket depth.
Width of Keratinized Tissue (KTW) | 6 months
  It is measured as the distance from the free gingival margin to the mucogingival junction, which will be measured at 6 months.
Wound Healing Index (WHI) | 3 months
  Early wound healing will be assessed semi-quantitatively with a composite index (Dastoor et al. 2007)designed to explore 4 areas/aspects of wound healing: i) the flap margin; ii) the interdental papilla; iii) the graft; and iv) the sutures. Weighted scores will be given to each parameter to develop a score designed to have a low value in a situation of perfect/uneventful early wound healing and higher values when aspects of wound failure will be detected
Root Coverage Aesthetic Score (Ref) | 6 months
  In order to assess the aesthetic outcome achieved after root coverage procedures, the Root Coverage Esthetic Score index (Cairo et al. 2009)will be used. This system evaluated 5 variables 6 months after the surgical procedure. The position of the gingival margin received 0, 3 or 6 points while all the other variables (marginal tissue contour, soft tissue texture, gingival color and MGJ alignment) were assigned either 0 or 1.

OTHER OUTCOMES:
Patient Concerns with Recession | 6 months
  This assessment is aimed at understanding the concerns that a patient has with recession of the gingival margin. The level of concern will be examined with a patient questionnaire on a 5-point Likert scale in terms of aesthetics, sensitivity to cold, sensitivity to brushing, root/tooth wear, fear to lose the involved teeth. The instrument will be used at baseline and at the 6-month follow-up appointment. The patient's response will be categorised based on their concern: 1)no concerned 2)a bit concerned 3)some concerned, 4)concerned 5)quite concerned
Time to recovery | 14 days
  A health diary, Periodontal Surgery Post-op (PSPostop), will be used to measure how the patient will be recovered following periodontal surgery. Each subject will be instructed to complete the diary each post-surgery day (PSD) for 14 days. A patient's daily response to each of the items will be categorized as 1) recovered defined as "no (1) or slight (2) trouble or discomfort" with that item or 2) substantial concern/ problem defined as "some, quite a bit or lots" as indicated by a response of 3 to 5 on the 5-point Likert-type scale

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Sanz, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Only on reasonable request to corresponding author

REFERENCES:
- [Background] Cairo F, Rotundo R, Miller PD, Pini Prato GP. Root coverage esthetic score: a system to evaluate the esthetic outcome of the treatment of gingival recession through evaluation of clinical cases. J Periodontol. 2009 Apr;80(4):705-10. doi: 10.1902/jop.2009.080565. PMID 19335093
- [Background] Dastoor SF, Travan S, Neiva RF, Rayburn LA, Giannobile WV, Wang HL. Effect of adjunctive systemic azithromycin with periodontal surgery in the treatment of chronic periodontitis in smokers: a pilot study. J Periodontol. 2007 Oct;78(10):1887-96. doi: 10.1902/jop.2007.070072. PMID 17915999
- [Background] Gobbato L, Nart J, Bressan E, Mazzocco F, Paniz G, Lops D. Patient morbidity and root coverage outcomes after the application of a subepithelial connective tissue graft in combination with a coronally advanced flap or via a tunneling technique: a randomized controlled clinical trial. Clin Oral Investig. 2016 Nov;20(8):2191-2202. doi: 10.1007/s00784-016-1721-7. Epub 2016 Jan 27. PMID 26814715
- [Background] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000
- [Background] Rebele SF, Zuhr O, Schneider D, Jung RE, Hurzeler MB. Tunnel technique with connective tissue graft versus coronally advanced flap with enamel matrix derivative for root coverage: a RCT using 3D digital measuring methods. Part II. Volumetric studies on healing dynamics and gingival dimensions. J Clin Periodontol. 2014 Jun;41(6):593-603. doi: 10.1111/jcpe.12254. PMID 24708338
- [Background] Zabalegui I, Sicilia A, Cambra J, Gil J, Sanz M. Treatment of multiple adjacent gingival recessions with the tunnel subepithelial connective tissue graft: a clinical report. Int J Periodontics Restorative Dent. 1999 Apr;19(2):199-206. PMID 10635186
- [Background] Zucchelli G, De Sanctis M. Long-term outcome following treatment of multiple Miller class I and II recession defects in esthetic areas of the mouth. J Periodontol. 2005 Dec;76(12):2286-92. doi: 10.1902/jop.2005.76.12.2286. PMID 16332241
- [Background] Zucchelli G, De Sanctis M. Treatment of multiple recession-type defects in patients with esthetic demands. J Periodontol. 2000 Sep;71(9):1506-14. doi: 10.1902/jop.2000.71.9.1506. PMID 11022782
- [Background] Zucchelli G, Mounssif I, Mazzotti C, Stefanini M, Marzadori M, Petracci E, Montebugnoli L. Coronally advanced flap with and without connective tissue graft for the treatment of multiple gingival recessions: a comparative short- and long-term controlled randomized clinical trial. J Clin Periodontol. 2014 Apr;41(4):396-403. doi: 10.1111/jcpe.12224. Epub 2014 Jan 22. PMID 24382170
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Background] Zuhr O, Rebele SF, Schneider D, Jung RE, Hurzeler MB. Tunnel technique with connective tissue graft versus coronally advanced flap with enamel matrix derivative for root coverage: a RCT using 3D digital measuring methods. Part I. Clinical and patient-centred outcomes. J Clin Periodontol. 2014 Jun;41(6):582-92. doi: 10.1111/jcpe.12178. Epub 2013 Nov 10. PMID 24117676
- [Derived] Gonzalez-Febles J, Romandini M, Laciar-Oudshoorn F, Noguerol F, Marruganti C, Bujaldon-Daza A, Zabalegui I, Sanz M. Tunnel vs. coronally advanced flap in combination with a connective tissue graft for the treatment of multiple gingival recessions: a multi-center randomized clinical trial. Clin Oral Investig. 2023 Jul;27(7):3627-3638. doi: 10.1007/s00784-023-04975-7. Epub 2023 Mar 29. PMID 36988824